CLINICAL TRIAL: NCT04096456
Title: Safety and Efficacy of Endoscopic Assisted Push Gastrostomy Using Gastropexy Technique
Brief Title: Safety and Efficacy of Endoscopic Assisted Push Gastrostomy Using Gastrostomy Technique
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: CHRISTUS Health (Other)
Collaborators: Baylor College of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: H-37260
Record Dates: First submitted 2019-09-18; First posted 2019-09-19 (Actual); Last update posted 2021-01-29 (Actual); Status verified 2021-01

CONDITIONS: Gastrostomy; Gastrostomy Complications; Gastrostomy Tube Site Complication; Pain, Postoperative
Keywords: Gastropexy; Endoscopic Gastropexy; Gastrostomy Tube
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Most pediatric gastroenterologists use an endoscopic pull technique to place gastrostomy tubes. We assessed an endoscopic gastropexy technique for gastrostomy tube placement that allows immediate placement of a low profile gastrostomy tube or gastro-jejunostomy tube. The procedure involves endoscopy with the placement of three T-fasteners that are placed through the skin into the stomach, placating and securing the stomach to the abdominal wall. This attachment process promotes formation of a stable gastrostomy tract, facilitating an immediate placement of a low profile gastrostomy button or gastro-jejunostomy tube. Serial dilators are then used to obtain the desired diameter of the ostomy for the tube placement. The gastropexy technique is most often associated with laparoscopic procedures involving gastric volvulus or complicated GERD, but little has been published investigating the outcomes of pediatric gastrostomy tube placement with the use of the gastropexy technique.

DETAILED DESCRIPTION:
This is a retrospective chart review. We will review charts of patients who underwent gastrostomy with gastropexy and primary percutaneous gastrostomy tube placement with pull through technique and compare immediate complications such as (pain, bleeding, and infection), and long term complications such as (feeding problems, pain, death, infection, bleeding and granulation), and for readmission in the 3 months following placement. Our control group will be the patients with primary percutaneous gastrostomy tube placement with pull through technique compared to the outcomes of the gastrostomy with gastropexy patients.

Inclusion Criteria:

Inclusion criteria is pediatric patients requiring an alternate means of nutrition with gastrostomy placement. Subjects ages 0-17 years of age. Data created starting 01/01/2005 to 07/31/2015.

Exclusion Criteria:

Patients that do not meet inclusion criteria.

Procedures: Most pediatric gastroenterologists use an endoscopic pull technique to place gastrostomy tubes. We will assess an endoscopic gastropexy technique for gastrostomy tube placement that allows immediate placement of a low profile gastrostomy tube or gastro-jejunostomy tube. The procedure involves endoscopy with the placement of three T-fasteners that are placed through the skin into the stomach, placating and securing the stomach to the abdominal wall. This attachment process promotes formation of a stable gastrostomy tract, facilitating an immediate placement of a low profile gastrostomy button or gastro-jejunostomy tube. Serial dilators are then used to obtain the desired diameter of the ostomy for the tube placement and a low profile gastrostomy button of appropriate size is placed. We will review complications both long term and short term of both the primary percutaneous gastrostomy tube placement with pull through technique compared to the outcomes of the gastrostomy with gastropexy patients.

Screening of GI cases at the Children's Hospital of San Antonio will be performed by PI and research staff to identify eligible patients. The subject record will be accessed and data recorded. The information recorded will be coded in the event a subject record requires subsequent reviews to obtain data. The subject record will be coded in order to protect subject PHI confidential. Please see section S for the data collection tool. The chart review will include records created starting 01/01/2005 - 06/26/2018.

Sample size: Local: 150, Worldwide: 150 The sample size is the any patient who underwent a gastrostomy with gastropexy or primary percutaneous gastrostomy tube placement with pull through technique by the gastroenterologists at the Children's Hospital of San Antonio.

Data Analysis: The primary comparison is the difference between immediate complications such as (pain, bleeding, and infection), and long term complications such as (feeding problems, pain, death, infection, bleeding and granulation) to evaluate efficacy and safety of gastrostomy with gastropexy.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria is pediatric patients requiring an alternate means of nutrition with gastrostomy placement. Subjects ages 0-17 years of age. Data created starting 01/01/2005 to 07/31/2015.

Exclusion Criteria:

* Patients that do not meet inclusion criteria.

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Retrospective chart review. The study population includes any patient who underwent a gastrostomy with gastropexy or primary percutaneous gastrostomy tube placement with pull through technique by the gastroenterologists at the Children's Hospital of San Antonio from 01/01/2005 - 06/26/2018.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2015-08-20 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Immediate and Long Term Complications | The retrospective chart review will include records created starting 01/01/2005 - 06/26/2018.
  The primary comparison is the difference between immediate complications such as (pain, bleeding, and infection), and long term complications such as (feeding problems, pain, death, infection, bleeding and granulation) to evaluate efficacy and safety of gastrostomy with gastropexy.

CONTACTS AND LOCATIONS:
Overall Officials: Javier Monagas, MD, Principal Investigator — The Children's Hospital of San Antonio
Locations (1):
- The Children's Hospital of San Antonio, San Antonio, Texas, United States